CLINICAL TRIAL: NCT05921201
Title: Preventing Depression of Chinese American Adolescents Through Mobile Health Application
Brief Title: Preventing Depression of Chinese American Adolescents by RRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Florida A&M University (Other); Florida State University (Other)
Responsible Party: Principal Investigator, Chieh Li, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NortheasternU-23-04-26
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Subclinical Depressive Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relax, Reflect, and Empower application (Experimental): Participants in the RRE group will select an Avatar from a pool of 20 Avatars as their companion over the 3 months. The Avatar wellness check-in in the RRE group includes a daily brief check-in of 5-minute/day (4 days/week), and a weekly full wellness check-in of 15 minutes/week for 3 months. The daily brief check-in includes a wellbeing and mood check and a 3-minute relaxation meditation. The weekly full wellness check-in includes reflection activities in addition to the daily check-in activities.
  Interventions: Behavioral: Relax, Reflect, and Empower mobile application
- Daily check-in text messages (Active Comparator): Participants will receive a wellness check-in text message 5 days/week [4 daily wellness check-in (2-3 minutes/day) +1 weekly wellness check-in (4-5 minutes/week)] for 3 months.
  Interventions: Behavioral: Relax, Reflect, and Empower mobile application

INTERVENTIONS:
Behavioral: Relax, Reflect, and Empower mobile application — Participants in the RRE group will select an Avatar from a pool of 20 Avatars as their companion over the 3 months. The Avatar wellness check-in in the RRE group includes a daily wellness check-in of 5-minute/day (4 days/week), and a weekly full wellness check-in of 15 minutes/week for 3 months. The daily brief check-in includes a wellbeing and mood check and a 3-minute relaxation meditation. The weekly full wellness check-in includes reflection activities in addition to the daily check-in activities.

SUMMARY:
The goal of this clinical trial is to test if a culturally sensitive mobile health application (Relax, Reflect, Empower-RRE) is feasible and effective in promoting psychological wellbeing and reducing depressive symptoms among Chinese American adolescents (CAA). We will conduct a pilot study of a community sample of 110 CAAs, ages 14-18. We will use adaptive randomization to assign 55 participants to the RRE intervention for 5 days/week for 3 months and 55 to the control group who will receive a wellness check-in text message 5 days/week for 3 months. The main aims/research questions are, 1) To evaluate feasibility and acceptability of RRE. Assessments include both subjective (CAAs' perceptions of feasibility and acceptability of RRE through Mobile Application Rating Scale and open-ended questions) and objective (CAAs' frequency and duration of RRE access automatically recorded) measures. Our hypothesis is that participants in the RRE group will find RRE feasible and acceptable. 2) To investigate CAAs' changes in depressive symptoms, coping self-efficacy, and psychological wellbeing. We will compare if these changes differ in the RRE group and control group. Participants in both RRE and control groups will complete measures of outcomes (depression, coping self-efficacy, psychological wellbeing) and influencing factors (acculturative stress, experiences of discrimination, life events) at three time points: baseline, the end of the preventive intervention (the12th week), and one-month after the intervention (the16th week). Our hypothesis is that CAAs in the RRE group will exhibit lower levels of depressive symptoms and higher levels of coping self-efficacy and psychological well-being in Weeks 12 and 16 than the baseline. Additionally, CAAs in the RRE group will exhibit greater improvement than the control group in the outcome measures from baseline to Weeks 12 and 16.

DETAILED DESCRIPTION:
Our clinical trial has two major aims. First, we will evaluate the feasibility and acceptability of RRE. Secondly, we will examine CAAs changes in depressive symptoms, coping self-efficacy, and psychological wellbeing, controlling for covariates (baseline, acculturative stress, experiences of discrimination, life events). As this project focuses on primary prevention for CAAs, we will use a community sample of 110 CAAs (based on power analyses and 20% attrition rate) in the Great Boston area, which ranks 5th metropolitan area with most Chinese Americans (n=277,312) in the U.S. The CAAs in this area are diverse in immigration history, socioeconomic status (SES), and parent education levels, which allows us to obtain representative participants from diverse socio-economic backgrounds and acculturation levels. The inclusion criteria for CAAs are (a) ethnic Chinese descent, born or grew up in the U.S, ages14 -18 enrolled in school, (b) understand and sign an informed consent (or assent for minors), and (c) have sixth grade reading level (to understand and complete proposed tasks).

Adaptive randomization (by gender, age, acculturation levels, SES, depression score) will be used to assign 55 participants to RRE for 5 days/week for 3 months and 55 to the control condition, who will receive a wellness check-in text message 5 days/week for 3 months. Participants in the RRE group will select an Avatar from a pool of 20 Avatars as their companion over the 3 months. The Avatar wellness check-in in the RRE group includes a daily brief check-in of 5-minute/day (4 days/week), and a weekly full wellness check-in of 15 minutes/week for 3 months. The daily brief check-in includes a wellbeing and mood check and a 3-minute relaxation meditation. The weekly full wellness check-in includes reflection activities in addition to the daily check-in activities. The reflection activities include 1) an innovative Ecomap to identify and quantify sources of stress and support, using a weighing scale, and 2) reflecting on existing and alternative coping strategies and their effectiveness. Avatar will introduce 3 different strategies and resources matching the key words/conditions from participant's responses from the pool of resources. The resources include evidence-based and culturally tailored self-help strategies, including Mindfulness Based Cognitive Therapy (MBCT) and Critical Consciousness (CC), and online and community mental health resources. For example, if a CAA girl seeks strategies to cope with bullying in school and her fear and anger, Avatar will present three relevant strategies from the tool bank of MBCT and CC, based on the key words she enters. The MBCT strategies will guide her how to cope with her feelings. The CC strategies will encourage her to examine systemic issues, stand up to bullying, and seek support. She can choose the strategies that she likes to try. Avatar will also present resources (online, school and community support) for her to consider. When the participant completes a daily or weekly wellness check-in, RRE will pop up the point/s earned toward monetary incentive/reward.

To ensure implementation fidelity of the prevention program and prevent attrition, Avatar will prompt each participant in the RRE group to do the wellness check-in daily. RRE will encourage CAAs to participate by showing the reward point/s earned each time completing a wellness check-in and the cumulated points for a monetary reward.

Staff from Florida Center for Interactive Media (FCIM) will resolve technical issues that may arise. To keep contact with participants in the control group, we will send them text messages five days per week, asking how they are doing, wishing them a nice day. Researchers will be monitoring the engagement activities in the RRE and control group daily.

ELIGIBILITY:
Inclusion Criteria: Participants must be CAAs (ethnic Chinese descent, born or grew up in the U.S) from the Greater Boston Area, Massachusetts, and meet the following inclusion criteria:

1. 14 -18 years old enrolled in school.
2. Understand and sign an informed consent (or assent for minors) document.
3. Sixth grade reading level (in order to understand and complete proposed tasks).

Exclusion Criteria:

1. Those who do not have sixth grade reading level to understand and complete the measures
2. Those who have a diagnosis of major depression or other mental disorders (that needs more extensive treatment than the Relax, Reflect, and Empower application -RRE program can provide)
3. Those who have a score of 3 or above in Patient Health Questionnaire-2 or Generalized Anxiety Disorder- 2 (who need more extensive treatment than the RRE program can provide)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | 2-5 minutes
  A 9-item valid, quick, and commonly used screening instrument for depression, It has demonstrated 90% of sensitivity and 78% of specificity in adolescents and is valid for Chinese American adolescents. Score ranges from 0 to 27. Scores 0 - 4 = No or Minimal depression. Higher scores indicate more severity of depression.

SECONDARY OUTCOMES:
Flourishing Scale | 5-7 minutes
  An 8-item measure of self-perceived success in relationships, self-esteem, purpose, and optimism. The measure has good psychometric properties and has been validated with Chinese and Chinese Americans. Score ranges from 8 to 56. Higher scores indicate more positive perception of oneself in important areas of functioning such as relationships, self-esteem, purpose, and optimism.
Coping self-efficacy scale (CSES) | 10 minutes
  CSES has 26 items with an 11-point scale for each item (with "Cannot do at all" = 0 at the lowest end, "Moderately certain can do" = 5 in the middle, and "Certain can do" =10 at the highest end of the scale. The CSES includes three factors: (a) problem-focused coping, (b) emotion-focused coping, and c) social support. CSES has demonstrated satisfactory reliability with culturally diverse adolescents. Higher scores represent higher self-reported abilities to cope with stressful circumstances.

CONTACTS AND LOCATIONS:
Overall Officials: Chieh Li, EdD, Principal Investigator — Northeastern University; Huijun Li, PhD, Principal Investigator — Florida A&M University; Shengli Dong, PhD, Principal Investigator — Florida State University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No